CLINICAL TRIAL: NCT04202965
Title: Open-label Study of PTG-300 in Subjects With Hereditary Hemochromatosis
Brief Title: PTG-300 in Subjects With Hereditary Hemochromatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTG-300-06
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2023-05

CONDITIONS: Hereditary Hemochromatosis
MeSH Terms: conditions — Hemochromatosis

STUDY DESIGN:
Intervention Model Description: Single Arm Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTG-300 (Experimental): PTG-300 Subcutaneous
  Interventions: Drug: PTG-300

INTERVENTIONS:
Drug: PTG-300 — Active treatment with PTG-300 injected subcutaneously.
  Other Names: Rusfertide

SUMMARY:
This study will be conducted at multiple sites and every patient will get treated with PTG-300. The objective of the study is to assess the effect of PTG-300 in treating adult hereditary hemochromatosis patients.

DETAILED DESCRIPTION:
This study is a multicenter, open-label study. The objective of the study is to assess the effect of PTG-300 on transferrin saturation (TSAT) and serum iron in adult hereditary hemochromatosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and older
* Confirmed diagnosis of HFE-related hereditary hemochromatosis with prior genotype testing
* Documented stable phlebotomy for ≥ 6 months
* Screening hemoglobin >11.5 g/dL
* Documented evidence of prior serum ferritin ≥500 ng/mL
* Serum ferritin >50 ng/mL and <300 ng/mL at screening

Exclusion Criteria:

* Clinically meaningful laboratory abnormality
* Receiving iron chelation therapy
* Receiving erythrocytapheresis
* Pregnant or lactating females
* Infection requiring hospitalization or intravenous antimicrobial therapy, or opportunistic infection within 3 months of dosing; any infections requiring antimicrobial therapy within 4 weeks of dosing.
* Serious or unstable medical or psychiatric condition that would prevent subject providing informed consent
* Organ damage from iron overload
* Primary or secondary immunodeficiency
* Positive hepatitis B or hepatitis C or known human immunodeficiency virus infection
* Known history of autoimmune/inflammatory diseases
* Any surgical procedures requiring general anesthesia within 1 month prior to screening or planned surgery during study
* History of invasive malignancies within last 2 years, except non-malignant skin cancer and local cured prostate cancer, cervical cancer, or ductal carcinoma in situ
* Receipt of an investigational agent within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - Protagonist Investigational Site, Fayetteville, Georgia
  - Protagonist Investigational Site, Bethesda, Maryland
  - Protagonist Investigational Site, Charlotte, North Carolina
  - Protagonist Investigational Site, Conroe, Texas
  - Protagonist Investigational Site, Dallas, Texas
  - Protagonist Investigational Site, Houston, Texas
  - Protagonist Investigational Site, Richmond, Virginia
  - Protagonist Investigational Site, Seattle, Washington
- Canada (2):
  - Protagonist Investigational Site, Halifax, Nova Scotia
  - Protagonist Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kowdley KV, Modi NB, Peltekian K, Vierling JM, Ferris C, Valone FH, Gupta S. Rusfertide for the treatment of iron overload in HFE-related haemochromatosis: an open-label, multicentre, proof-of-concept phase 2 trial. Lancet Gastroenterol Hepatol. 2023 Dec;8(12):1118-1128. doi: 10.1016/S2468-1253(23)00250-9. Epub 2023 Oct 17. PMID 37863080

RESULTS

PARTICIPANT FLOW:
Groups:
- PTG-300: PTG-300 injected subcutaneously. PTG-300 doses individually titrated with doses ranging from 10 mg to 40 mg once weekly or twice a week.
Period: Overall Study
Arm/Group | PTG-300
Started | 16
Completed | 12
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Did not meet inclusion criteria | 1

BASELINE CHARACTERISTICS:
Groups:
- PTG-300: PTG-300: Active treatment with PTG-300 subcutaneously
Arm/Group | PTG-300
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (3.87)

OUTCOME MEASURES:

1. Primary Outcome: Effect of PTG-300 on Transferrin Saturation
Description: Change from Baseline to Week 24 (or End of Treatment) in transferrin saturation (TSAT) as measured by blood laboratory tests.
Time Frame: Week 24 (or End of Treatment if treated for less than 24 weeks)
Population: Subjects who had paired values to allow determination of change from baseline
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | PTG-300
Number analyzed (Participants) | 14
percent saturation | -6.07 (19.4)

2. Primary Outcome: Effect of PTG-300 on Serum Iron
Description: Change from Baseline to Week 24 (or End of Treatment) in serum iron as measured by blood laboratory tests.
Time Frame: Week 24 (or End of Treatment if treated for less than 24 weeks)
Population: Subjects who had paired values to allow determination of change from baseline
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | PTG-300
Number analyzed (Participants) | 14
micromol/L | -2.34 (9.76)

3. Secondary Outcome: Effect of PTG-300 on Phlebotomy Frequency
Description: Change in number of phlebotomies in 24-weeks before treatment compared with the number of phlebotomies during 24-weeks of treatment with PTG-300.
Time Frame: Over 24 weeks
Population: Enrolled population
Measure: Mean (Standard Deviation); unit: phlebotomies/week
Arm/Group | PTG-300
Number analyzed (Participants) | 16
phlebotomies/week | 0.00 (0.01)

4. Other Pre Specified Outcome: Mental Component Summary of SF-36
Description: Change from Baseline to Week 24 (or End of Treatment) in Mental Component Summary of the SF-36.
  The SF-36 is a questionnaire of health status based on 36 questions distributed into eight domains of daily life that are frequently evaluated as influenced by disease. Values in each domain range from 0 to 100, with higher scores indicating better health condition. A summary measure, Mental Component Summary (MCS), for mental health can be calculated. The MCS ranges from 0 (low functioning) to 100 (high functioning).
Time Frame: Week 24 (or End of Treatment if treated for less than 24 weeks)
Population: Subjects who have a Score at Baseline and at Week 24 or End of Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTG-300
Number analyzed (Participants) | 15
units on a scale | -0.251 (9.379)

5. Other Pre Specified Outcome: Physical Component Summary of SF-36
Description: Change from Baseline to Week 24 (or End of Treatment) in Physical Component Summary of the SF-36.
  The SF-36 is a questionnaire of health status based on 36 questions distributed into eight domains of daily life that are frequently evaluated as influenced by disease. Values in each domain range from 0 to 100, with higher scores indicating better health condition. A summary measure, Physical Component Summary (PCS), for mental health can be calculated. The PCS ranges from 0 (low functioning) to 100 (high functioning).
Time Frame: Week 24 (or End of Treatment if treated for less than 24 weeks)
Population: Subjects who have a Score at Baseline and at Week 24 or End of Treatment
Measure: Mean (Standard Deviation); unit: units on a scake
Arm/Group | PTG-300
Number analyzed (Participants) | 15
units on a scake | 2.263 (6.528)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Safety was assessed using the National Institutes of Health (NIH) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria.
Arm/Group | PTG-300
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTG-300 (N=16)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Pre-existing condition diagnosed during study. Not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PTG-300 (N=16)
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Fatigue (General disorders) | 2
Inflammation (General disorders) | 1
Injection site bruising (General disorders) | 1
Injection site discomfort (General disorders) | 1
Injection site erythema (General disorders) | 2
Injection site haematoma (General disorders) | 1
Injection site haemorrhage (General disorders) | 1
Injection site induration (General disorders) | 1
Injection site pain (General disorders) | 5
Injection site pruritus (General disorders) | 3
Injection site swelling (General disorders) | 1
Malaise (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Gastrointestinal bacterial overgrowth (Infections and infestations) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04202965/Prot_SAP_000.pdf